CLINICAL TRIAL: NCT06107400
Title: Study to Evaluate the Safety and Efficacy of RM-004 Cells for the Treatment of Hemoglobin H-Constant Spring Disease
Brief Title: Safety and Efficacy of RM-004 Cells for Hemoglobin H-Constant Spring Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army (Other)
Collaborators: Guangzhou Reforgene Medicine Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-RM-004-01
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-10

CONDITIONS: Alpha Thalassemia Hemoglobin H Constant Spring; Hemoglobinopathies; Hereditary Diseases
Keywords: RM-004; Hemoglobin H-Constant Spring disease; Alpha-Thalassemia; Gene therapy; CBE
MeSH Terms: conditions — Hemoglobinopathies; Genetic Diseases, Inborn; alpha-Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RM-004 (Experimental): RM-004 (ex vivo gene-edited CD34+ autologous hematopoietic stem cells) will be administered as a single intravenous infusion
  Interventions: Genetic: RM-004

INTERVENTIONS:
Genetic: RM-004 — Intravenous infusion of gene-edited CD34+autologous hematopoietic stem cells (RM-004) after myeloablative conditioning with busulfan.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of RM-004 for Hemoglobin H-Constant Spring disease.

DETAILED DESCRIPTION:
This is a non-randomized, one-arm, open label study to evaluate the safety and efficacy of RM-004 for autologous hematopoietic stem cell transplantation (HSCT) for the treatment of Hemoglobin H-Constant Spring disease. Five subjects aged from 12 to 35 years will be recruited in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign informed consent by themselves or their legal guardians and complete the study procedures, follow-up examination and treatment.
2. At the time of screening, subjects should be aged from 12 to 35 years old, regardless of gender.
3. History of at least 100 mL/kilograms (kg)/year of packed red blood cells (pRBC) transfusions in the prior 2 years before screening.
4. Subjects diagnosed with Hemoglobin H-Constant Spring disease (--/ααCS) with HBA2 c.427T>C mutation.

Exclusion Criteria:

1. Subject who has an available HLA-matched/well-matched HSCT donor for allogeneic hematopoietic stem cell transplantation (HSCT).
2. Prior HSCT or gene therapy.
3. History of severe hemorrhagic disease.
4. Clinically significant active bacterial, viral, fungal or parasitic infections per investigator's judgement at the time of screening.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with engraftment | Within 42 days after RM-004 infusion
  Proportion of subjects with successful neutrophil engraftment (first day of 3 consecutive measurements of absolute neutrophil count [ANC] ≥0.5×10^9/L on 3 different days) after RM-004 infusion.
Safety of RM-004 infusion | From signing of informed consent up to 24 months after RM-004 infusion
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs)
Proportion of subjects who achieve transfusion independence | Up to 24 months after RM-004 infusion
  Transfusion independence (TI) was defined as a weighted average hemoglobin (Hb) ≥ 9 g/dL without any red blood cells transfusions for a continuous period of ≥12 months at any time during the study after RM-004 infusion.

SECONDARY OUTCOMES:
Incidence of all-cause mortality | From signing of informed consent up to 24 months after RM-004 infusion
  Incidence of all-cause mortality
Proportion of subjects who stop receiveing transfusion ≥ 6 months | Up to 24 months after RM-004 infusion
  Proportion of subjects who stop receiveing transfusion ≥ 6 months
Duration of transfusion independence | Up to 24 months after RM-004 infusion
  Duration of TI was calculated as the time from the start of TI up to the last available Hb at which the TI criteria are still met. Time period of TI will start when subjects achieve a Hb ≥ 9 g/dL with no transfusions in the preceding 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Zhang, MD, Principal Investigator — The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army
Locations (1):
- The 923rd Hospital of Joint Logistics Support Force of People's Liberation Army, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No